CLINICAL TRIAL: NCT02440373
Title: Plasma Cytochrome c as Biomarker of Traumatic Injury and Predictor of Outcome
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Rosalind Franklin University of Medicine and Science (Other)
Responsible Party: Sponsor
Other Study IDs: AHC IRB# 5458
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2018-03

CONDITIONS: Trauma; Blunt Injury; Blunt Trauma; Accident; Multiorgan Injury
MeSH Terms: conditions — Wounds and Injuries; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood drawn within 15 minutes of arrival to the Emergency Department and at 24, 48, and 74 hours. Each sample will be processed and stored for subsequent analysis of cytochrome c and other markers of mitochondrial injury that may become available at a later time.
Oversight: Data Monitoring Committee: No

SUMMARY:
Cytochrome c is a mitochondrial protein that plays a key role in energy metabolism. When mitochondria are injured, cytochrome c may leave mitochondria and reach the bloodstream. The investigators plan to investigate whether circulating cytochrome c levels may serve as biomarker of traumatic injury correlating with (1) severity of traumatic injury, (2) development of organ dysfunction, and (3) clinical outcomes. The Trauma Services at ALGH will enroll over 8 months 100 consecutive trauma patients who require intubation for mechanical ventilation and survive to hospital admission. The Resuscitation Institute at RFUMS will measure cytochrome c levels in plasma taken upon hospital admission and subsequently at 24, 48, and 72 hours, with additional plasma stored for markers to be defined at a later time. Blood cytochrome c levels will be analyzed in relation to severity of traumatic injury, development of organ dysfunction, and clinical outcomes including survival and functional status (adjusted for covariates such as age, gender, type of trauma, time to stabilization, comorbidities, etc.) using information obtained as part of routine medical care. Successful completion of this project will support blood cytochrome c as biomarker of traumatic injury which could be used to identify severity, predict outcomes, and assess novel mitochondrial protective strategies.

DETAILED DESCRIPTION:
The investigators propose to determine whether plasma cytochrome c could serve as clinical biomarker of traumatic injury by examining the relationship between plasma levels of cytochrome c and the severity of the initial injury upon arrival to the hospital, subsequent development of organ dysfunction, and clinical outcomes. Cytochrome c is a mitochondrial protein that plays a crucial role in energy metabolism enabling transfer of electrons from complex III (i.e., cytochrome c reductase) to complex IV (cytochrome c oxidase). Upon mitochondrial injury and contingent on severity, cytochrome c may be released to the cytosol and subsequently to the bloodstream. The rationale for this project stems from: (1) observations at the Resuscitation Institute in animal models of cardiac arrest and resuscitation in which plasma cytochrome c correlates directly with the severity of post-resuscitation left ventricular dysfunction and inversely with survival and (2) observations by others reporting a correlation between plasma cytochrome c and severity of organ injury. The investigators hypothesize that plasma cytochrome c measured upon arrival to the hospital reflects the severity of the initial traumatic injury resulting from the aggregate effects of direct injury to organs, ischemic injury consequent to blood loss, delays in stabilization, and preexistent comorbidity - all factors that can injure mitochondria. The investigators further hypothesize that the initial cytochrome c plasma level combined with the levels measured during the subsequent three days of hospitalization correlate with the development of organ dysfunction, and clinical outcomes. The current proposal is structured in three specific aims:

Specific Aim 1 (collection of blood samples and clinical data): For this aim the investigator plans to enroll 100 consecutive trauma victims admitted to Advocate Lutheran General Hospital (ALGH) over a period of 8 months presenting with single or multisystem injuries and meeting specific entry and exclusion criteria developed to ensure a broad range of injury severity. Blood will be sampled within 15 minutes of hospital arrival (e.g., in the Emergency Department or Operating Room) and subsequently at 24, 48, and 72 hours. Plasma will be separated and stored at -80 °C for subsequent batch measurement of cytochrome c (and other markers of mitochondrial injury that may become available at the time of analysis) in the Resuscitation Institute at Rosalind Franklin Univer-sity of Medicine and Science (RFUMS). Clinical data will be extracted from tools used clinically - including the Illinois Trauma Registry Worksheet and the medical record - and used to: (i) record severity of initial traumatic injury by calculating the Trauma Score - Injury Severity Score (TRISS) along with a detailed assessment of individual organs injury; (ii) estimate the severity of blood loss based on base deficit and transfusion needs; (iii) determine subsequent development of organ dysfunction by calculating the Multiple Organ Dysfunction Score (MODS) and the Sequential Organ Failure Score; and (iv) assess outcomes by measuring length of stay in the Intensive Care Unit (ICU), length of stay in the hospital, survival upon hospital discharge, and functional status upon hospital discharge.

Specific Aim 2 (analysis of plasma cytochrome c): Frozen samples of arterial plasma, stored at -80°C at ALGH, will be transferred to the Resuscitation Institute at RFU and cytochrome c measured using electrochemiluminescence.

Specific Aim 3 (statistical analysis and modeling): A database devoid of patient identifiers will be created merging the clinical information with values of plasma cytochrome c levels and other markers as they become available. Considering the pilot nature of the project, statistical modeling and analysis will be primarily exploratory focused on identifying relationships between plasma cytochrome c levels upon hospital arrival and clinical elements contributing of the severity of primary traumatic injury. The analysis and modeling will also include examining the predictive value of the initial and subsequent plasma cytochrome c levels on development of organ dysfunction and clinical outcomes.

The long-term goal of the project is to develop plasma cytochrome c as biomarker of traumatic injury and other clinical conditions associated with mitochondrial injury that could be used at the bedside - i.e., after developing point of care assays - for (1) assessing severity of illness, (2) prognostication of outcome, and (3) clinical re-search on novel therapeutic interventions aimed at reducing mitochondrial injury.

ELIGIBILITY:
Inclusion criteria:

Age 18 years or older. Blunt mechanism for the primary injury. Time from injury to hospital arrival is ≤ 2 hours Mechanical ventilation for any reason, including surgery, within the initial 24 hours from hospital arrival.

Any one of the following:

* Systolic blood pressure <90 mmHg (Class III shock- >30 %blood loss) within 4 hours from hospital arrival.
* Base deficit > 4 mmol/l in the first blood gas upon hospital arrival
* Transfusion of ≥ 2 units of packed red blood cells within ≤12 hours from hospital arrival.

Exclusion Criteria (ANY SINGLE ONE):

Known disease with life expectancy <6 months. Penetrating mechanism for the primary injury. Death within 4 hours from hospital arrival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of both genders suffering acute non-penetrating traumatic injury.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Plasma cytochrome c levels in relation to severity of traumatic injury | Day one.
  Relationship between plasma levels of cytochrome c and the initial severity of traumatic injury as assessed by the TRISS and the severity of initial presentation based on transfusion requirements and (if available) by blood gas and chemistry analysis along with lactic acid.

SECONDARY OUTCOMES:
Plasma cytochrome c levels in relation to development of organ dysfunction and hospital outcomes | From hospital admission until the date of discharge from the hospital, up to 26 weeks.
  Relationship between plasma levels of cytochrome c and subsequent development of organ dysfunction assessed by daily measurements of MODS and SOFA and various clinical outcomes including length of stay in ICU and in the hospital, survival to hospital discharge, and functional status upon discharge.
Individual organ contribution to plasma cytochrome c levels | From hospital admission until the date of the last cytochrome c measurement (i.e., day three from hospital admission).
  Contribution of individual organs injured to plasma cytochrome c levels (e.g., liver injury is likely to produce greater mitochondrial injury that thoracic injury given the greater mitochondrial density in liver tissue).

CONTACTS AND LOCATIONS:
Overall Officials: Raul Gazmuri, MD, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

REFERENCES:
- [Background] Bertini I, Cavallaro G, Rosato A. Cytochrome c: occurrence and functions. Chem Rev. 2006 Jan;106(1):90-115. doi: 10.1021/cr050241v. No abstract available. PMID 16402772
- [Background] Giege P, Grienenberger JM, Bonnard G. Cytochrome c biogenesis in mitochondria. Mitochondrion. 2008 Jan;8(1):61-73. doi: 10.1016/j.mito.2007.10.001. Epub 2007 Oct 11. PMID 18033741
- [Background] Radhakrishnan J, Wang S, Ayoub IM, Kolarova JD, Levine RF, Gazmuri RJ. Circulating levels of cytochrome c after resuscitation from cardiac arrest: a marker of mitochondrial injury and predictor of survival. Am J Physiol Heart Circ Physiol. 2007 Feb;292(2):H767-75. doi: 10.1152/ajpheart.00468.2006. Epub 2006 Oct 13. PMID 17040974
- [Background] Ow YP, Green DR, Hao Z, Mak TW. Cytochrome c: functions beyond respiration. Nat Rev Mol Cell Biol. 2008 Jul;9(7):532-42. doi: 10.1038/nrm2434. PMID 18568041
- [Background] Radhakrishnan J, Kolarova JD, Ayoub IM, Gazmuri RJ. AVE4454B--a novel sodium-hydrogen exchanger isoform-1 inhibitor--compared less effective than cariporide for resuscitation from cardiac arrest. Transl Res. 2011 Feb;157(2):71-80. doi: 10.1016/j.trsl.2010.11.004. Epub 2010 Dec 15. PMID 21256459
- [Background] Alleyne T, Joseph J, Sampson V. Cytochrome-c detection: a diagnostic marker for myocardial infarction. Appl Biochem Biotechnol. 2001 Feb;90(2):97-105. doi: 10.1385/abab:90:2:97. PMID 11297391
- [Background] Renz A, Burek C, Mier W, Mozoluk M, Schulze-Osthoff K, Los M. Cytochrome c is rapidly extruded from apoptotic cells and detectable in serum of anticancer-drug treated tumor patients. Adv Exp Med Biol. 2001;495:331-4. doi: 10.1007/978-1-4615-0685-0_46. No abstract available. PMID 11774588
- [Background] Adachi N, Hirota M, Hamaguchi M, Okamoto K, Watanabe K, Endo F. Serum cytochrome c level as a prognostic indicator in patients with systemic inflammatory response syndrome. Clin Chim Acta. 2004 Apr;342(1-2):127-36. doi: 10.1016/j.cccn.2003.12.011. PMID 15026273
- [Background] Barczyk K, Kreuter M, Pryjma J, Booy EP, Maddika S, Ghavami S, Berdel WE, Roth J, Los M. Serum cytochrome c indicates in vivo apoptosis and can serve as a prognostic marker during cancer therapy. Int J Cancer. 2005 Aug 20;116(2):167-73. doi: 10.1002/ijc.21037. PMID 15800951
- [Background] Hosoya M, Nunoi H, Aoyama M, Kawasaki Y, Suzuki H. Cytochrome c and tumor necrosis factor-alpha values in serum and cerebrospinal fluid of patients with influenza-associated encephalopathy. Pediatr Infect Dis J. 2005 May;24(5):467-70. doi: 10.1097/01.inf.0000160995.07461.b8. PMID 15876954
- [Background] Hosoya M, Kawasaki Y, Katayose M, Sakuma H, Watanabe M, Igarashi E, Aoyama M, Nunoi H, Suzuki H. Prognostic predictive values of serum cytochrome c, cytokines, and other laboratory measurements in acute encephalopathy with multiple organ failure. Arch Dis Child. 2006 Jun;91(6):469-72. doi: 10.1136/adc.2005.078436. Epub 2006 Jan 27. PMID 16443616
- [Background] Sakaida I, Kimura T, Yamasaki T, Fukumoto Y, Watanabe K, Aoyama M, Okita K. Cytochrome c is a possible new marker for fulminant hepatitis in humans. J Gastroenterol. 2005 Feb;40(2):179-85. doi: 10.1007/s00535-004-1517-4. PMID 15770402
- [Background] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228
- [Background] Cook R, Cook D, Tilley J, Lee K, Marshall J; Canadian Critical Care Trials Group. Multiple organ dysfunction: baseline and serial component scores. Crit Care Med. 2001 Nov;29(11):2046-50. doi: 10.1097/00003246-200111000-00002. PMID 11700393
- [Background] Jacobs S, Zuleika M, Mphansa T. The Multiple Organ Dysfunction Score as a descriptor of patient outcome in septic shock compared with two other scoring systems. Crit Care Med. 1999 Apr;27(4):741-4. doi: 10.1097/00003246-199904000-00027. PMID 10321663
- [Background] Peres Bota D, Melot C, Lopes Ferreira F, Nguyen Ba V, Vincent JL. The Multiple Organ Dysfunction Score (MODS) versus the Sequential Organ Failure Assessment (SOFA) score in outcome prediction. Intensive Care Med. 2002 Nov;28(11):1619-24. doi: 10.1007/s00134-002-1491-3. Epub 2002 Sep 6. PMID 12415450
- [Background] Raedler C, Voelckel WG, Wenzel V, Krismer AC, Schmittinger CA, Herff H, Mayr VD, Stadlbauer KH, Lindner KH, Konigsrainer A. Treatment of uncontrolled hemorrhagic shock after liver trauma: fatal effects of fluid resuscitation versus improved outcome after vasopressin. Anesth Analg. 2004 Jun;98(6):1759-1766. doi: 10.1213/01.ANE.0000117150.29361.5A. PMID 15155342
- [Background] Voelckel WG, Convertino VA, Lurie KG, Karlbauer A, Schochl H, Lindner KH, Trimmel H. Vasopressin for hemorrhagic shock management: revisiting the potential value in civilian and combat casualty care. J Trauma. 2010 Jul;69 Suppl 1:S69-74. doi: 10.1097/TA.0b013e3181e44937. PMID 20622623
- [Background] Anand T, Skinner R. Arginine vasopressin: the future of pressure-support resuscitation in hemorrhagic shock. J Surg Res. 2012 Nov;178(1):321-9. doi: 10.1016/j.jss.2012.02.062. Epub 2012 Mar 17. PMID 22480832
- [Background] Davis DP, Garberson LA, Andrusiek DL, Hostler D, Daya M, Pirrallo R, Craig A, Stephens S, Larsen J, Drum AF, Fowler R. A descriptive analysis of Emergency Medical Service Systems participating in the Resuscitation Outcomes Consortium (ROC) network. Prehosp Emerg Care. 2007 Oct-Dec;11(4):369-82. doi: 10.1080/10903120701537147. PMID 17907019
- [Background] Morley P. Steady as a ROC: the Resuscitation Outcomes Consortium. Resuscitation. 2008 Aug;78(2):105-6. doi: 10.1016/j.resuscitation.2008.06.007. No abstract available. PMID 18620110
- [Background] Atkins DL, Everson-Stewart S, Sears GK, Daya M, Osmond MH, Warden CR, Berg RA; Resuscitation Outcomes Consortium Investigators. Epidemiology and outcomes from out-of-hospital cardiac arrest in children: the Resuscitation Outcomes Consortium Epistry-Cardiac Arrest. Circulation. 2009 Mar 24;119(11):1484-91. doi: 10.1161/CIRCULATIONAHA.108.802678. Epub 2009 Mar 9. PMID 19273724
- [Background] Newgard CD, Schmicker RH, Hedges JR, Trickett JP, Davis DP, Bulger EM, Aufderheide TP, Minei JP, Hata JS, Gubler KD, Brown TB, Yelle JD, Bardarson B, Nichol G; Resuscitation Outcomes Consortium Investigators. Emergency medical services intervals and survival in trauma: assessment of the "golden hour" in a North American prospective cohort. Ann Emerg Med. 2010 Mar;55(3):235-246.e4. doi: 10.1016/j.annemergmed.2009.07.024. Epub 2009 Sep 23. PMID 19783323
- [Background] Bulger EM, May S, Kerby JD, Emerson S, Stiell IG, Schreiber MA, Brasel KJ, Tisherman SA, Coimbra R, Rizoli S, Minei JP, Hata JS, Sopko G, Evans DC, Hoyt DB; ROC investigators. Out-of-hospital hypertonic resuscitation after traumatic hypovolemic shock: a randomized, placebo controlled trial. Ann Surg. 2011 Mar;253(3):431-41. doi: 10.1097/SLA.0b013e3181fcdb22. PMID 21178763
- [Background] Bulger EM, Guffey D, Guyette FX, MacDonald RD, Brasel K, Kerby JD, Minei JP, Warden C, Rizoli S, Morrison LJ, Nichol G; Resuscitation Outcomes Consortium Investigators. Impact of prehospital mode of transport after severe injury: a multicenter evaluation from the Resuscitation Outcomes Consortium. J Trauma Acute Care Surg. 2012 Mar;72(3):567-73; discussion 573-5; quiz 803. doi: 10.1097/TA.0b013e31824baddf. PMID 22491538
- [Background] Arnold DM, Burns KE, Adhikari NK, Kho ME, Meade MO, Cook DJ; McMaster Critical Care Interest Group. The design and interpretation of pilot trials in clinical research in critical care. Crit Care Med. 2009 Jan;37(1 Suppl):S69-74. doi: 10.1097/CCM.0b013e3181920e33. PMID 19104228
- [Background] Ashe D, Alleyne T, Iwuoha E. Serum cytochrome c detection using a cytochrome c oxidase biosensor. Biotechnol Appl Biochem. 2007 Apr;46(Pt 4):185-9. doi: 10.1042/BA20060103. PMID 17059389
- [Background] Li X, Liu H, He X, Song Z. Determination of cytochrome c in human serum and pharmaceutical injections using flow injection chemiluminescence. Appl Biochem Biotechnol. 2010 Feb;160(4):1065-73. doi: 10.1007/s12010-009-8598-8. Epub 2009 Apr 4. PMID 19347266
- [Background] Yan S, Xu X, Sheng Y, Sun H, Wu J, Tang L. Disposable biosensor based on Au nanoparticles-modified CdS nanorod arrays for detection cytochrome c. J Nanosci Nanotechnol. 2011 Dec;11(12):10320-3. doi: 10.1166/jnn.2011.5012. PMID 22408904
- [Background] Ayoub IM, Kolarova JD, Kantola RL, Radhakrishnan J, Wang S, Gazmuri RJ. Zoniporide preserves left ventricular compliance during ventricular fibrillation and minimizes postresuscitation myocardial dysfunction through benefits on energy metabolism. Crit Care Med. 2007 Oct;35(10):2329-36. doi: 10.1097/01.ccm.0000280569.87413.74. PMID 17944021
- [Background] Gazmuri RJ, Radhakrishnan J. Protecting mitochondrial bioenergetic function during resuscitation from cardiac arrest. Crit Care Clin. 2012 Apr;28(2):245-70. doi: 10.1016/j.ccc.2012.02.001. PMID 22433486
- [Background] Cairns CB, Moore FA, Haenel JB, Gallea BL, Ortner JP, Rose SJ, Moore EE. Evidence for early supply independent mitochondrial dysfunction in patients developing multiple organ failure after trauma. J Trauma. 1997 Mar;42(3):532-6. doi: 10.1097/00005373-199703000-00023. PMID 9095123
- [Background] Ott M, Robertson JD, Gogvadze V, Zhivotovsky B, Orrenius S. Cytochrome c release from mitochondria proceeds by a two-step process. Proc Natl Acad Sci U S A. 2002 Feb 5;99(3):1259-63. doi: 10.1073/pnas.241655498. Epub 2002 Jan 29. PMID 11818574
- [Background] von Harsdorf R, Li PF, Dietz R. Signaling pathways in reactive oxygen species-induced cardiomyocyte apoptosis. Circulation. 1999 Jun 8;99(22):2934-41. doi: 10.1161/01.cir.99.22.2934. PMID 10359739
- [Background] Petrosillo G, Ruggiero FM, Pistolese M, Paradies G. Ca2+-induced reactive oxygen species production promotes cytochrome c release from rat liver mitochondria via mitochondrial permeability transition (MPT)-dependent and MPT-independent mechanisms: role of cardiolipin. J Biol Chem. 2004 Dec 17;279(51):53103-8. doi: 10.1074/jbc.M407500200. Epub 2004 Oct 8. PMID 15475362
- [Background] de Moissac D, Gurevich RM, Zheng H, Singal PK, Kirshenbaum LA. Caspase activation and mitochondrial cytochrome C release during hypoxia-mediated apoptosis of adult ventricular myocytes. J Mol Cell Cardiol. 2000 Jan;32(1):53-63. doi: 10.1006/jmcc.1999.1057. PMID 10652190
- [Background] Loor G, Kondapalli J, Iwase H, Chandel NS, Waypa GB, Guzy RD, Vanden Hoek TL, Schumacker PT. Mitochondrial oxidant stress triggers cell death in simulated ischemia-reperfusion. Biochim Biophys Acta. 2011 Jul;1813(7):1382-94. doi: 10.1016/j.bbamcr.2010.12.008. Epub 2010 Dec 23. PMID 21185334
- [Background] Li P, Nijhawan D, Budihardjo I, Srinivasula SM, Ahmad M, Alnemri ES, Wang X. Cytochrome c and dATP-dependent formation of Apaf-1/caspase-9 complex initiates an apoptotic protease cascade. Cell. 1997 Nov 14;91(4):479-89. doi: 10.1016/s0092-8674(00)80434-1. PMID 9390557
- [Background] Budihardjo I, Oliver H, Lutter M, Luo X, Wang X. Biochemical pathways of caspase activation during apoptosis. Annu Rev Cell Dev Biol. 1999;15:269-90. doi: 10.1146/annurev.cellbio.15.1.269. PMID 10611963
- [Background] Saleh A, Srinivasula SM, Acharya S, Fishel R, Alnemri ES. Cytochrome c and dATP-mediated oligomerization of Apaf-1 is a prerequisite for procaspase-9 activation. J Biol Chem. 1999 Jun 18;274(25):17941-5. doi: 10.1074/jbc.274.25.17941. PMID 10364241
- [Background] Zou H, Li Y, Liu X, Wang X. An APAF-1.cytochrome c multimeric complex is a functional apoptosome that activates procaspase-9. J Biol Chem. 1999 Apr 23;274(17):11549-56. doi: 10.1074/jbc.274.17.11549. PMID 10206961
- [Background] Zager RA, Johnson AC, Hanson SY. Proximal tubular cytochrome c efflux: determinant, and potential marker, of mitochondrial injury. Kidney Int. 2004 Jun;65(6):2123-34. doi: 10.1111/j.1523-1755.2004.00638.x. PMID 15149325
- [Background] Osaka A, Hasegawa H, Tsuruda K, Inokuchi N, Yanagihara K, Yamada Y, Aoyama M, Sawada T, Kamihira S. Serum cytochrome c to indicate the extent of ongoing tumor cell death. Int J Lab Hematol. 2009 Jun;31(3):307-14. doi: 10.1111/j.1751-553X.2008.01033.x. Epub 2008 Feb 12. PMID 18279425
- [Background] Liu X, Xie W, Liu P, Duan M, Jia Z, Li W, Xu J. Mechanism of the cardioprotection of rhEPO pretreatment on suppressing the inflammatory response in ischemia-reperfusion. Life Sci. 2006 Apr 4;78(19):2255-64. doi: 10.1016/j.lfs.2005.09.053. Epub 2005 Dec 5. PMID 16336978
- [Background] Marenzi G, Giorgio M, Trinei M, Moltrasio M, Ravagnani P, Cardinale D, Ciceri F, Cavallero A, Veglia F, Fiorentini C, Cipolla CM, Bartorelli AL, Pelicci P. Circulating cytochrome c as potential biomarker of impaired reperfusion in ST-segment elevation acute myocardial infarction. Am J Cardiol. 2010 Nov 15;106(10):1443-9. doi: 10.1016/j.amjcard.2010.07.014. Epub 2010 Sep 23. PMID 21059434
- [Background] Narula J, Pandey P, Arbustini E, Haider N, Narula N, Kolodgie FD, Dal Bello B, Semigran MJ, Bielsa-Masdeu A, Dec GW, Israels S, Ballester M, Virmani R, Saxena S, Kharbanda S. Apoptosis in heart failure: release of cytochrome c from mitochondria and activation of caspase-3 in human cardiomyopathy. Proc Natl Acad Sci U S A. 1999 Jul 6;96(14):8144-9. doi: 10.1073/pnas.96.14.8144. PMID 10393962
- [Background] Radhakrishnan J, Ayoub IM, Gazmuri RJ. Activation of caspase-3 may not contribute to postresuscitation myocardial dysfunction. Am J Physiol Heart Circ Physiol. 2009 Apr;296(4):H1164-74. doi: 10.1152/ajpheart.00338.2008. Epub 2009 Feb 20. PMID 19234092
- [Background] Narula J, Arbustini E, Chandrashekhar Y, Schwaiger M. Apoptosis and the systolic dysfunction in congestive heart failure. Story of apoptosis interruptus and zombie myocytes. Cardiol Clin. 2001 Feb;19(1):113-26. doi: 10.1016/s0733-8651(05)70198-3. PMID 11787805
- [Background] Communal C, Sumandea M, de Tombe P, Narula J, Solaro RJ, Hajjar RJ. Functional consequences of caspase activation in cardiac myocytes. Proc Natl Acad Sci U S A. 2002 Apr 30;99(9):6252-6. doi: 10.1073/pnas.092022999. Epub 2002 Apr 23. PMID 11972044
- [Background] Pettila V, Pettila M, Sarna S, Voutilainen P, Takkunen O. Comparison of multiple organ dysfunction scores in the prediction of hospital mortality in the critically ill. Crit Care Med. 2002 Aug;30(8):1705-11. doi: 10.1097/00003246-200208000-00005. PMID 12163780
- [Background] Durham RM, Moran JJ, Mazuski JE, Shapiro MJ, Baue AE, Flint LM. Multiple organ failure in trauma patients. J Trauma. 2003 Oct;55(4):608-16. doi: 10.1097/01.TA.0000092378.10660.D1. PMID 14566110
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239